CLINICAL TRIAL: NCT06843278
Title: Donor Breast Milk and Serum Ferritin Levels in Very Preterm Infants: A Prospective, Observational Study
Brief Title: Donor Breast Milk and Serum Ferritin Levels in Very Preterm Infants
Status: Completed | Type: Observational
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Other Study IDs: 1878559
Record Dates: First submitted 2025-02-20; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-01

CONDITIONS: Ferritin Levels in Very Preterm Infants
Keywords: Breast milk; Donor breast milk; Ferritin level; very preterm infants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Very preterm infants receiving breast milk
  Interventions: Other: maternal breast milk
- Very preterm infants receiving donor breast milk
  Interventions: Other: Donor breast milk

INTERVENTIONS:
Other: maternal breast milk — Very preterm infants receiving maternal breast milk
  Groups: Very preterm infants receiving breast milk
Other: Donor breast milk — Very preterm infants receiving donor breast milk
  Groups: Very preterm infants receiving donor breast milk

SUMMARY:
This study compares the iron levels in very preterm infants receiving donor breast (DBM) milk to very preterm infants receiving maternal breast milk (MBM).

ELIGIBILITY:
Inclusion Criteria:

1. All preterm infants born between 29 weeks and 0 days -32 weeks and 6 days of gestational age and admitted to the NICU at Advent Health for Children
2. Received either MBM or DBM starting between 5 to10 days of life

   a. Infants receiving >50% feeding volume by DBM for the first 14 days of life will be considered to have received predominantly DBM. The comparison group will be infants who received > 50% of MBM for the first 14 days of life.
3. Parent able to read and write in the English language.

Exclusion Criteria:

1. Death prior to completion of participation
2. Extremis with likelihood of death prior to completion of participation in the study
3. Blood transfusion as determined by clinical team during the study
4. Major congenital anomaly or genetic syndrome and
5. Major surgical GI conditions that preclude feeding

Ages: 2 Weeks to 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Very preterm infants
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
The Average Serum ferritin level in very preterm infants | Until four weeks of age or discharge
  The average serum ferritin level (ng/ml) in very preterm infants receiving donor breast milk or maternal breast milk

SECONDARY OUTCOMES:
The Average Hemoglobin levels (g/dl) in very preterm infants | Until four weeks of age or discharge
  The average Hemoglobin levels (g/dL) in very preterm infants receiving donor breast milk or maternal breast milk
The Average Bilirubin Levels (mg/dL) in very preterm infants | until four weeks of age or discharge
  The average Hemoglobin levels (g/dL) in very preterm infants receiving donor breast milk or maternal breast milk

CONTACTS AND LOCATIONS:
Overall Officials: Anoop Pulickal, MD, Principal Investigator — AdvenHealth
Locations (1):
- AdventHealth, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gao C, Miller J, Middleton PF, Huang YC, McPhee AJ, Gibson RA. Changes to breast milk fatty acid composition during storage, handling and processing: A systematic review. Prostaglandins Leukot Essent Fatty Acids. 2019 Jul;146:1-10. doi: 10.1016/j.plefa.2019.04.008. Epub 2019 May 1. PMID 31186148
- [Background] Maisels MJ, Gifford K. Breast-feeding, weight loss, and jaundice. J Pediatr. 1983 Jan;102(1):117-8. doi: 10.1016/s0022-3476(83)80305-9. No abstract available. PMID 6848709
- [Background] Joy R, Krishnamurthy S, Bethou A, Rajappa M, Ananthanarayanan PH, Bhat BV. Early versus late enteral prophylactic iron supplementation in preterm very low birth weight infants: a randomised controlled trial. Arch Dis Child Fetal Neonatal Ed. 2014 Mar;99(2):F105-9. doi: 10.1136/archdischild-2013-304650. Epub 2013 Dec 3. PMID 24302687
- [Background] Kc A, Rana N, Malqvist M, Jarawka Ranneberg L, Subedi K, Andersson O. Effects of Delayed Umbilical Cord Clamping vs Early Clamping on Anemia in Infants at 8 and 12 Months: A Randomized Clinical Trial. JAMA Pediatr. 2017 Mar 1;171(3):264-270. doi: 10.1001/jamapediatrics.2016.3971. PMID 28114607
- [Background] Mercer JS, Erickson-Owens DA, Deoni SCL, Dean DC 3rd, Collins J, Parker AB, Wang M, Joelson S, Mercer EN, Padbury JF. Effects of Delayed Cord Clamping on 4-Month Ferritin Levels, Brain Myelin Content, and Neurodevelopment: A Randomized Controlled Trial. J Pediatr. 2018 Dec;203:266-272.e2. doi: 10.1016/j.jpeds.2018.06.006. Epub 2018 Jul 6. PMID 30473033
- [Background] German KR, Vu PT, Comstock BA, Ohls RK, Heagerty PJ, Mayock DE, Georgieff M, Rao R, Juul SE; PENUT Consortium. Enteral Iron Supplementation in Infants Born Extremely Preterm and its Positive Correlation with Neurodevelopment; Post Hoc Analysis of the Preterm Erythropoietin Neuroprotection Trial Randomized Controlled Trial. J Pediatr. 2021 Nov;238:102-109.e8. doi: 10.1016/j.jpeds.2021.07.019. Epub 2021 Jul 27. PMID 34324880
- [Background] Taufek NM, Cartwright D, Hewavitharana A, Koorts P, McConachy H, Shaw N, Whitfield K, Davies M. TO INVESTIGATE THE EFFECT OF THE PASTEURISATION PROCESS ON TRACE ELEMENTS IN DONOR BREAST MILK. Arch Dis Child. 2016 Sep;101(9):e2. doi: 10.1136/archdischild-2016-311535.27. PMID 27540206
- [Background] Mohd-Taufek N, Cartwright D, Davies M, Hewavitharana AK, Koorts P, McConachy H, Shaw PN, Sumner R, Whitfield K. The effect of pasteurization on trace elements in donor breast milk. J Perinatol. 2016 Oct;36(10):897-900. doi: 10.1038/jp.2016.88. Epub 2016 Jun 2. PMID 27253894
- [Background] Mannel R, Peck JD. Outcomes Associated With Type of Milk Supplementation Among Late Preterm Infants. J Obstet Gynecol Neonatal Nurs. 2018 Jul;47(4):571-582. doi: 10.1016/j.jogn.2017.11.005. Epub 2017 Dec 27. PMID 29287170
- [Background] Stoltz Sjostrom E, Ohlund I, Tornevi A, Domellof M. Intake and macronutrient content of human milk given to extremely preterm infants. J Hum Lact. 2014 Nov;30(4):442-9. doi: 10.1177/0890334414546354. Epub 2014 Aug 12. PMID 25117506
- [Background] Hard AL, Nilsson AK, Lund AM, Hansen-Pupp I, Smith LEH, Hellstrom A. Review shows that donor milk does not promote the growth and development of preterm infants as well as maternal milk. Acta Paediatr. 2019 Jun;108(6):998-1007. doi: 10.1111/apa.14702. Epub 2019 Jan 25. PMID 30565323
- [Background] Quigley M, Embleton ND, McGuire W. Formula versus donor breast milk for feeding preterm or low birth weight infants. Cochrane Database Syst Rev. 2019 Jul 19;7(7):CD002971. doi: 10.1002/14651858.CD002971.pub5. PMID 31322731
- [Background] Arslanoglu S, Ziegler EE, Moro GE; World Association of Perinatal Medicine Working Group On Nutrition. Donor human milk in preterm infant feeding: evidence and recommendations. J Perinat Med. 2010 Jul;38(4):347-51. doi: 10.1515/jpm.2010.064. PMID 20443660
- [Background] American Academy of Pediatrics Policy Statement. Breastfeeding and the use of breast milk. Pediatrics 2012; 129:e827-841